CLINICAL TRIAL: NCT06828952
Title: Risk Factors of Failure of Conservative Treatment in Acute Non Complicated Appendicitis
Acronym: appendicitis
Status: Not yet recruiting | Type: Observational
Sponsor: Ahmed Mohammed Hussein Sayed (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Ahmed Mohammed Hussein Sayed, Principal investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: acute appendicitis
Record Dates: First submitted 2024-12-04; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-12

CONDITIONS: Conservative Management
Keywords: Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Ceftriaxone; Metronidazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- (1) Male or female patients é diagnosis of acute appendicitis.: Patients who presented with complaints of right lower quadrant pain with symptoms and signs strongly suggestive of uncomplicated acute appendicitis that was confirmed on ultrasonography, were included. The modified Alvarado score and adult appendicitis score were calculated.
  Interventions: Drug: ceftriaxone; Drug: ceftriaxone 1 gm/12 hourly and IV metronidazole 500 mg/8 hourly

INTERVENTIONS:
Drug: ceftriaxone — ceftriaxone 1 gm/12 hourly and IV metronidazole 500 mg/8 hourly
Drug: ceftriaxone 1 gm/12 hourly and IV metronidazole 500 mg/8 hourly — Conservative management

SUMMARY:
From this study, it can be concluded that patients who meet the following criteria are more likely to fail expectant management and thus should not be considered for the NOM of uncomplicated acute appendicitis. These include the duration of symptoms before presenting to a surgical emergency , the presence of fever within 24 hours of presenting to a surgical emergency, TLC cells/dL, CRP mg/L, appendix diameter mm, modified Alvarado score , and adult appendicitis score .

DETAILED DESCRIPTION:
Expectant management with intravenous antibiotic therapy alone has emerged as an effective alternative to appendectomy for the treatment of uncomplicated acute appendicitis . It is important to identify patients at the onset of the disease who are likely to have successful outcomes for conservative management.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients é diagnosis of acute appendicitis .
* Patients with ages: from 16 to 60 years old.

Exclusion Criteria:

* complicated AA (appendicolith, perforation, peri appendicular abscess or suspicion of a tumor).
* inflammatory bowel disease.
* inability to co-operate and give informed consent.
* diffuse peritonitis.
* antibiotic documented allergy & allergy to contrast media .
* Patients with serious comorbid conditions DM & renal insufficiency, serum creatinine > 150 μmol/l .
* Pregnant & lactating patient.
* Patients with bleeding diathesis and those on anticoagulants.
* Patients with advanced malignancies & patient on immunosuppressive drugs .
* Patients with previous appendectomy.
* Extreme of age.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Male or female patients é diagnosis of acute appendicitis Patients with ages: from 16 to 60 years old
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-22 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-02 (Estimated)

PRIMARY OUTCOMES:
Risk factors of failure of conservative treatment in acute non complicated appendicitis | One year
  modified Alvarado score and adult appendicitis score

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Shindoh J, Niwa H, Kawai K, Ohata K, Ishihara Y, Takabayashi N, Kobayashi R, Hiramatsu T. Predictive factors for negative outcomes in initial non-operative management of suspected appendicitis. J Gastrointest Surg. 2010 Feb;14(2):309-14. doi: 10.1007/s11605-009-1094-1. PMID 19936849
- [Background] Hansson J, Khorram-Manesh A, Alwindawe A, Lundholm K. A model to select patients who may benefit from antibiotic therapy as the first line treatment of acute appendicitis at high probability. J Gastrointest Surg. 2014 May;18(5):961-7. doi: 10.1007/s11605-013-2413-0. Epub 2013 Nov 22. PMID 24263678
- [Background] Walker C, Moosavi A, Young K, Fluck M, Torres D, Widom K, Wild J. Factors Associated with Failure of Nonoperative Management for Complicated Appendicitis. Am Surg. 2019 Aug 1;85(8):865-870. PMID 31560305
- [Background] Loftus TJ, Brakenridge SC, Croft CA, Stephen Smith R, Efron PA, Moore FA, Mohr AM, Jordan JR. Successful nonoperative management of uncomplicated appendicitis: predictors and outcomes. J Surg Res. 2018 Feb;222:212-218.e2. doi: 10.1016/j.jss.2017.10.006. Epub 2017 Nov 13. PMID 29146455
- [Background] Cervellin G, Mora R, Ticinesi A, Meschi T, Comelli I, Catena F, Lippi G. Epidemiology and outcomes of acute abdominal pain in a large urban Emergency Department: retrospective analysis of 5,340 cases. Ann Transl Med. 2016 Oct;4(19):362. doi: 10.21037/atm.2016.09.10. PMID 27826565
- See also: include the duration of symptoms before presenting to a surgical emergency , the presence of fever within 24 hours of presenting to a surgical emergency, TLC cells/dL, CRP mg/L, appendix diameter mm, modified Alvarado score , and adult appendicitis scor — https://pubmed.ncbi.nlm.nih.gov/19936849/